CLINICAL TRIAL: NCT05019924
Title: An Exploratory Investigation of Dietary Supplementation and the Effect on Common PMS and Menstrual Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semaine Health (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20216
Record Dates: First submitted 2021-08-10; First posted 2021-08-25 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Menstrual Pain; Menstrual Discomfort
Keywords: PMS; Menstrual symptoms
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Dietary supplement
  Interventions: Dietary Supplement: Semaine
- Control arm (No Intervention): No intervention given

INTERVENTIONS:
Dietary Supplement: Semaine — The dietary supplement is designed, and marketed commercially to be taken in servings of two capsules per day, up to four times per day (a total of 8 capsules daily). Most consumers, however, will only take a serving three times per day, or one with each major meal (breakfast, lunch and dinner).
  Arms: Intervention arm

SUMMARY:
Dietary supplementation is widely used to alleviate various symptoms of PMS and menstruation such as bloating and cramping. Providing a combination of synergistic dietary supplements is hypothesized to significantly reduce self-reported PMS and menstrual discomfort when compared with a baseline without the intervention.

DETAILED DESCRIPTION:
This is an open-label observational trial to study the effectiveness of a commercial dietary supplement and its effect on common symptoms of normal menstrual discomfort.

It is hypothesized that the dietary supplement marketed as Semaine PMS & Period Support will improve subjective wellbeing and biomarkers in trial participants.

A total of 58 participants will be recruited for the trial following screening, with the expectation that at least 51 will complete the trial. The trial will be fully remote, and all participants will undergo a menstrual cycle without intervention to establish a baseline, and then will be given the intervention (dietary supplement) for a second menstrual cycle. For both menstrual cycles the participants will complete a subjective wellbeing survey and provide a blood sample for biomarker analysis.

The biomarker analysis will be performed through an at-home fingerprick blood test. To maximize consistency, the tests should be performed on the same days of each cycle - preferably on days 4 or 5. If absolutely necessary, however one day of buffer on either side will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Female, aged 18-40
* Willingness to refrain from ibuprofen or naproxen sodium (such as Advil, Aleve, Motrin or Midol) during each period (pill bleed) during the study
* Ability to take oral medication and be willing to adhere to the dietary supplement regimen
* Use of hormonal contraception for at least 3 months prior to screening and agreement to use such a method during study participation. Hormonal contraception must allow for pill bleeds to occur.
* Moderate self-reported discomfort during menstruation related to bloating, pelvic cramps, fatigue or mood swings. On a scale of 1-10, participants must report at least a 4 on two or more symptoms.
* Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

* Current use of GnRH agonists and antagonists including Lupron or Orilissa
* Current use of an extended activity hormonal contraception (for example, Depo-provera or Nexplanon)
* Current use of hyperthyroid medication such as methimazole
* Current use of blood thinning medication
* Pregnancy, lactation, or attempting to become pregnant during study
* Known allergic reactions to components of the dietary supplement (sunflower oil, ashwagandha, curcumin, resveratrol, Boswellia, milk thistle, quercetin or catechins)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in perceived discomfort associated with menstruation [Time Frame: Baseline to 8 weeks) | 8 week intervention period
  Perceived discomfort caused by several of the most common menstrual symptoms Cramping Bloating Gastrointestinal issues (diarrhea or constipation) Feeling tired Feeling down emotionally Feeling anxious Headache
  Each endpoint will be reported by the participant on a scale of perceived discomfort at the end of each menstrual cycle. Participants will complete the surveys for each menstrual cycle. The study uses a questionnaire including a scale from 0-7 to assess the severity of symptoms(0=no symptoms and 7=very severe symptoms).
  To ensure consistency between participants, each survey will be completed on days 7 or 8 after they stop hormonal contraception usage (or begin placebo pills).

SECONDARY OUTCOMES:
Change in blood biomarkers: C-Reactive Protein (CRP) and 25-hydroxyvitamin D [Time Frame: Baseline to 8 weeks] | 8 week intervention period
  Change in C-Reactive Protein (CRP) and 25-hydroxyvitamin D biomarkers measured with an at-home blood test after 8 weeks compared to baseline results.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study will be conducted in accordance with the following publication and data sharing policies: the study will be published in an open-access preprint server, and every attempt will be made to publish the results in an open-access peer-reviewed journal. The study administrators (CitrusLabs) will be acknowledged in the publications. This trial will be registered with clinicaltrials.gov and results will be submitted to clinicaltrials.gov following publication.